CLINICAL TRIAL: NCT06767969
Title: Effect of Acetaminophen on Neurological Outcome in Acute Ischemic Stroke Patients Undergoing Endovascular Treatment
Acronym: ACEAIS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Ruquan Han, Dr, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: wxy20241217ACEAIS
Record Dates: First submitted 2025-01-06; First posted 2025-01-10 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-02

CONDITIONS: Ischemic Stroke
Keywords: ischemic stroke; Endovascular treatments; acetaminophen
MeSH Terms: conditions — Ischemic Stroke | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (No Intervention): There was no intervention and it was performed according to standardized clinical management
- Acetaminophen group (Experimental): Acetaminophenl 500mg (500mg/50ml) was infused intravenously every 6 hours( a single infusion is completed within 15-30 minutes) from the beginning of endovascular treatment to 48 hours after treatment.
  Interventions: Drug: Acetaminophen

INTERVENTIONS:
Drug: Acetaminophen — Acetaminophenl 500mg (500mg/50ml) was infused intravenously every 6 hours( a single infusion is completed within 15-30 minutes) from the beginning of endovascular treatment to 48 hours after treatment.
  Arms: Acetaminophen group

SUMMARY:
Neuro-inflammation response plays an important role in the development of acute ischemic stroke(AIS). The aim of this study was to conduct a prospective randomized controlled study on the effect of acetaminophen on long-term neurological prognosis in AIS patients undergoing endovascular treatment(EVT). The primary outcome was the incidence of neurological independence (mRS 0-2, modified Rankin scale) at 90 days after surgery. The secondary outcome measures were early neurological outcome (NIHSS score at 7 days after surgery or at discharge) and the incidence of symptomatic intracerebral hemorrhage during hospitalization. This study explored the effect of acetaminophen on the prognosis of neurological function of patients, and the expected results provide evidence of safety and effectiveness for acetaminophen to improve the prognosis of neurological function of patients, and provide theoretical and practical basis for the subsequent "new use of old drugs" of acetaminophen and large sample and multi-center clinical research or clinical application.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old; computer tomography angiogram (CTA), Magnetic Resonance Angiography (MRA), MRA) or digital subtraction angiography (DSA) confirmed the presence of large intracranial artery occlusion (intracranial internal carotid artery, anterior cerebral artery, M1 and M2 segments of middle cerebral artery, basilar artery, posterior cerebral artery); Endovascular treatment including intra-arterial thrombolysis, mechanical thrombectomy, angioplasty, etc. was performed (within 24 hours of onset). The NIHSS score at admission was 6-26. The mRS Score before onset was less than 2. Patients or their legal representatives provided written informed consent

Exclusion Criteria:

The mRS Score before the stroke was ≥2. Intracranial hemorrhagic diseases: cerebral hemorrhage, subarachnoid hemorrhage, etc. Patients had a history of coagulopathy, systemic bleeding, thrombocytopenia or neutropenia. Renal insufficiency with elevated serum creatinine (> 2 times the upper limit of normal); Severe hepatic insufficiency or liver disease, with elevations in liver enzymes (aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase, or gamma-glutamyl transpeptidase) of more than twice the upper limit of the normal range; Patients with severe active liver disease; Patients with severe heart and lung diseases considered by the investigator to be ineligible for the study; DSA examination is contraindicated, severe contrast agent allergy or iodine contrast agent is absolutely contraindicated; Women of childbearing age, pregnant or lactating women who have a negative pregnancy test but refuse to use effective contraception; Inability to complete the study due to mental disorders, cognitive or emotional disorders; Allergy to acetaminophen; Other patients who were not included in the study in the opinion of the investigator (reasons indicated)

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 892 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
The incidence of functional independence | 90 (±7) days after treatment
  modified Rankin score from 0 to 2

IPD SHARING:
Plan to Share IPD: Undecided
Patient privacy data were involved